CLINICAL TRIAL: NCT03446729
Title: Enhancing Memory to Facilitate Weight Loss: Tracking, Recording and Coaching
Acronym: TRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kerri Boutelle, Professor, Pediatrics and Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 131518
Record Dates: First submitted 2018-02-08; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory Self Monitoring (MSM) (Experimental): Intervention: Guided self-help Behavioral Weight Loss. The MSM group is assigned to self-monitor in "habit books" what they consume in their previous meal immediately prior to each meal, similar to other studies exploring the effect of episodic meal memory on food intake.
  Interventions: Behavioral: Guided Self-Help Behavioral Weight Loss
- Caloric Self Monitoring (CSM) (Active Comparator): Intervention: Guided self-help Behavioral Weight Loss. The CSM group is assigned to self-monitor what food they consume, and the associated caloric content after each meal in their "habit books" in line with traditional BWL self-monitoring.
  Interventions: Behavioral: Guided Self-Help Behavioral Weight Loss

INTERVENTIONS:
Behavioral: Guided Self-Help Behavioral Weight Loss — Guided self-help Behavioral Weight Loss including 7 visits over 12 weeks. The treatment content includes self-monitoring, healthy eating, stimulus control, increasing physical activity, reducing sedentary activity, planning ahead for high-risk situations, and relapse prevention. The 7 visits are conducted with a behavioral coach to give participants educational materials and to promote accountability. The behavioral coach's role in the gshBWL program is to measure participant weight, collect self-monitoring booklets, clarify materials, and problem-solve barriers to adherence.
  Other Names: gshBWL

SUMMARY:
The objective of this application is to pilot test and evaluate the acceptability and efficacy of a program to facilitate weight loss by enhancing memory for a recently consumed meal.

DETAILED DESCRIPTION:
Once enrolled, all participants will receive behavioral weight loss treatment. Treatment will be 12 weeks in duration and will consist of 7 sessions. The content of sessions will provide the main elements described in behavioral therapy programs for obesity, based on empirical literature. Participants will be provided handouts, and the handout content will be based on our clinic treatment manual and published behavior therapy protocols. The program will be administered in individual 30-60-min sessions with a behavioral coach meeting every other week. This program emphasizes self-monitoring of food intake. It also emphasizes gradual weight loss, increasing physical activity, and improving diet through permanent lifestyle changes. Program topics include: self-monitoring of eating behavior, physical activity, changing the home environment and nutrition education. All treatment sessions will be conducted by licensed clinical health psychologists or psychology doctoral level students with experience in leading weight loss interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be overweight (BMI between 25-40)
2. Participant must be between the ages of 18-55
3. Participant can read at a minimum of an 5th grade level in English
4. Participant is willing to participate and to commit to 12 weeks of treatment and attendance at assessments

Exclusion Criteria:

1. Participant is unable to exercise (ex., due to physical or medical reasons)
2. Major psychiatric disorder diagnoses, including an eating disorder
3. Diagnoses of a serious current physical disease (such as diabetes) for which physician supervision of diet is needed
4. Participant who takes medications that would influence weight and eating, or cognitive functioning, such as attention, concentration, or mental status

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2015-12-03 (Actual)

PRIMARY OUTCOMES:
Attendance | Post-Treatment (12 weeks following baseline)
  The number of treatment visits attended
Attrition | Change from baseline at an average of 12 weeks
  The percentage of participant attrition from each treatment arm
Self-Monitoring Adherence | Post-Treatment (12 weeks following baseline)
  The number of days that participants self-monitor
Acceptability | Measured at an average of 12 weeks following baseline
  Average of likert ratings of self-monitoring method, was it "easier," "more helpful," or "more convenient" than any methods participants may have used to self-monitor in the past
Weight Change | Change from baseline at an average of 12 weeks and 24 weeks
  Weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Working Memory | Change from baseline at an average of 12 weeks and 24 weeks
  Digit Span: scaled total forward and backward score
Food specific memory | Change from baseline at an average of 12 weeks and 24 weeks
  A food version of the California Verbal Learning Test. Sum of words recalled across the five recall trials of list A (high calorie food, low calorie food, neutral words) as a measure of global index of verbal learning ability.

OTHER OUTCOMES:
Restraint | Change from baseline at an average of 12 weeks and 24 weeks
  Restraint subscale from the Three Factor Eating Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, PhD, Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robinson E, Aveyard P, Daley A, Jolly K, Lewis A, Lycett D, Higgs S. Eating attentively: a systematic review and meta-analysis of the effect of food intake memory and awareness on eating. Am J Clin Nutr. 2013 Apr;97(4):728-42. doi: 10.3945/ajcn.112.045245. Epub 2013 Feb 27. PMID 23446890